CLINICAL TRIAL: NCT00482209
Title: Study of 400mcg Versus 800mcg Buccal Misoprostol Following Mifepristone 200mg for Abortion up to 63 Days Gestation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Dr. Beverly Winikoff, Gynuity Health Projects
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1.1.6
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2009-10-12 (Estimated); Status verified 2009-10

CONDITIONS: Induced Abortion
Keywords: mifepristone, misoprostol, medical abortion
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- 1 (Active Comparator): 200mg mifepristone followed by 400mcg misoprostol
  Interventions: Drug: Mifepristone, misoprostol
- 2 (Active Comparator): 200mg mifepristone followed by 800mcg misoprostol
  Interventions: Drug: mifepristone, misoprostol

INTERVENTIONS:
Drug: Mifepristone, misoprostol — 200mg mifepristone followed by 400mcg misoprostol 36-48 hours later
  Arms: 1
Drug: mifepristone, misoprostol — 200mg mifepristone followed by 800mcg misoprostol 36-48 hours later
  Arms: 2

SUMMARY:
This double-blind, randomized study will compare the efficacy and acceptability of mifepristone 200mg followed in 36-48 hours by 400mcg or 800mcg of buccal misoprostol (i.e., in the cheeks) for termination of pregnancy in women up to 63 days LMP.

DETAILED DESCRIPTION:
The goal of this study is to provide answers to the following four questions:

1. Is a regimen of medical abortion with mifepristone using 400mcg buccal misoprostol as effective and acceptable as using 800mcg buccal misoprostol up to 63 days since the last menstrual period (LMP)?
2. Are the side effects with buccal use tolerable for women?
3. Is buccal administration of misoprostol acceptable to women?
4. When given a choice, do women prefer to take misoprostol at home or in the clinic?

ELIGIBILITY:
Inclusion Criteria:

* Women 18 years or over presenting for abortion services who consent to participate
* good general health
* assessed by a clinician to have an intrauterine pregnancy less than 64 days LMP on Study Day 1 and to be eligible for medical abortion
* Have ready access to a telephone and emergency transportation;
* Be willing to provide an address and/or telephone number for purposes of follow-up

Exclusion Criteria:

* Conditions which contraindicate the use of mifepristone or misoprostol
* Women presenting for medical abortion who do not consent to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1220 (Estimated)
Dates: Start 2007-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Need for surgical completion for ongoing viable pregnancies at follow up visit (Study day 12-15) or for incomplete abortion at extended follow up visit (Study day (19-22). | Study day 12-15 for ongoing viable pregnancies or Study day 19-22 for incomplete abortion at extended follow up visit

SECONDARY OUTCOMES:
Side-effects, acceptability for women | side effects and acceptability recorded at exit interview

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Erica Chong, MPH, Study Director — Gynuity Health Projects; Tamuna Tsereteli, MD, MSc, PhD, Study Director — Gynuity Health Projects
Locations (4):
- Georgia (3):
  - Maternity House #2, Tbilisi
  - Maternity House #4, Tbilisi
  - Zhordania Institute of Human Reproduction, Tbilisi
- Hocmon Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- See also: Related Info — http://www.gynuity.org